CLINICAL TRIAL: NCT00160602
Title: A Phase III Multi-center, Double-blind, Placebo-controlled, Parallel Group 24-Week Study to Assess the Efficacy and Safety of Two Dose Regimens of Liquid Certolizumab Pegol as Additional Medication to Methotrexate in the Treatment of Signs and Symptoms of Rheumatoid Arthritis and in Prevention of Joint Damage in Patients With Active Rheumatoid Arthritis Who Have an Incomplete Response to Methotrexate.
Brief Title: A Study of Liquid Certolizumab Pegol as Additional Medication to Methotrexate in the Treatment of Signs and Symptoms of Rheumatoid Arthritis and in Prevention of Joint Damage in Patients With Active Rheumatoid Arthritis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: UCB Pharma (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: C87050; EudraCT Number: 2005-002326-63
Record Dates: First submitted 2005-09-08; First posted 2005-09-12 (Estimated); Last update posted 2020-12-01 (Actual); Status verified 2020-11

CONDITIONS: Rheumatoid Arthritis
Keywords: Rheumatoid Arthritis; Certolizumab Pegol, Cimzia
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Certolizumab Pegol

INTERVENTIONS:
Drug: Certolizumab Pegol

SUMMARY:
A 24 week study in which patients are given study medication and assessed for signs and symptoms of rheumatoid arthritis. X-rays are performed to assess the progress of joint damage during the study.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be at least 18 years old at the screening visit.
* Patients must have a diagnosis of adult-onset RA of at least six months duration but not longer than fifteen years as defined by the 1987 American College of Rheumatology classification criteria.
* Patients must have active RA disease as defined by:

  * 9 tender joints at Screening and Baseline.
  * 9 swollen joints at Screening and Baseline. and fulfilling 1 of the following 2 criteria during the screening period:
  * 30 mm/hour ESR (Westergren), or CRP >15 mg/L.
* Patients must have received treatment with MTX (with or without folic acid) for at least 6 months prior to the Baseline visit. The dose of MTX and route of administration must have been stable for at least 2 months prior to the baseline visit. The minimum stable dose of MTX allowed is 10 mg weekly.
* Patients must be willing to complete an X-ray of the hands and feet 24 weeks after randomization even if they are no longer receiving study treatment in the present study, provided they have not withdrawn their informed consent.

Exclusion Criteria:

* Patients must not have a diagnosis of any other inflammatory arthritis (e.g., psoriatic arthritis or ankylosing spondylitis).
* Patients must not have a secondary, non-inflammatory type of arthritis (e.g. OA or fibromyalgia)
* Female patients who are breast feeding, pregnant, or plan to become pregnant during the trial or for three months following last dose of study drug.
* Patients with a history of tuberculosis or positive chest X-ray for tuberculosis or positive
* Patients at a high risk of infection (e.g. leg ulcers, indwelling urinary catheter and persistent or recurrent chest infections and patients who are permanently bed ridden or wheelchair bound).
* Patients with known human immunodeficiency virus (HIV) infection.
* Patients with an active malignancy of any type or a history of malignancy (except basal cell carcinoma of the skin that has been excised prior to study start).
* Patients with a current or recent history, as determined by the Investigator, of severe, progressive, and/or uncontrolled renal, hepatic, hematological, gastrointestinal, endocrine, pulmonary, cardiac, neurological, or cerebral disease which would interfere with the patient's participation in the trial.
* Patients with a history of, or suspected, demyelinating disease of the central nervous system (e.g. multiple sclerosis or optic neuritis).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 590
Dates: Start 2005-06; Primary Completion 2006-09 (Actual); Study Completion 2006-09 (Actual)

PRIMARY OUTCOMES:
Compare efficacy of two dose regimens of certolizumab pegol in combination with MTX to MTX alone in patients with RA measured by the ACR20 at week 24.

SECONDARY OUTCOMES:
Assess Safety and Tolerability of two dose regimens of certolizumab pegol in combination with MTX and MTX alone in patients with RA; prevention of joint damage in patients with RA; Health Outcomes Measures

CONTACTS AND LOCATIONS:
Overall Officials: UCB Clinical Trial Call Center, Study Director — UCB Pharma
Locations (70):
- United States (17):
  - Montgomery, Alabama
  - Sun City West, Arizona
  - Palm Desert, California
  - Pasadena, California
  - Santa Maria, California
  - Naples, Florida
  - Palm Harbor, Florida
  - South Miami, Florida
  - New Orleans, Louisiana
  - St Louis, Missouri
  - New Brunswick, New Jersey
  - Stratford, New Jersey
  - New York, New York
  - Rochester, New York
  - Canfield, Ohio
  - Wynnewood, Pennsylvania
  - San Antonio, Texas
- Bulgaria (3):
  - Pleven
  - Sofia
  - Stara Zagora
- Chile (2):
  - Santiago
  - Temuco
- Rijeka, Croatia
- Czechia (7):
  - Brno
  - Hlučín
  - Ostrava-Poruba
  - Prague
  - Sokolov
  - UherskeHradiste
  - Zlín
- Tallinn, Estonia
- Israel (7):
  - Afula
  - Ashkelon
  - Beer Yaakov
  - Haifa
  - Jerusalem
  - Ramat Gan
  - Rehovot
- Latvia (2):
  - Daugavpils
  - Riga
- Lithuania (5):
  - Alytus
  - Kaunas
  - Klaipėda
  - Panevezys
  - Šiauliai
- Mexico (5):
  - D. F.
  - Mexicalli
  - México
  - Monterrey
  - Tijuana
- Poland (6):
  - Bialystok
  - Elblag
  - Krakow
  - Lublin
  - Sopot
  - Torun
- Russia (3):
  - Moscow
  - Saint Petersburg
  - Yaroslavl
- Serbia (3):
  - Belgrade
  - Niška Banja
  - Novi Sad
- Slovakia (2):
  - Košice
  - Piešťany
- Ukraine (6):
  - Dnipro
  - Donetsk
  - Ivano-Frankivsk
  - Kiev
  - Simferopol
  - Zaporizhzhya

REFERENCES:
- [Result] Smolen J, Landewe RB, Mease P, Brzezicki J, Mason D, Luijtens K, van Vollenhoven RF, Kavanaugh A, Schiff M, Burmester GR, Strand V, Vencovsky J, van der Heijde D. Efficacy and safety of certolizumab pegol plus methotrexate in active rheumatoid arthritis: the RAPID 2 study. A randomised controlled trial. Ann Rheum Dis. 2009 Jun;68(6):797-804. doi: 10.1136/ard.2008.101659. Epub 2008 Nov 17. PMID 19015207
- [Result] Strand V, Smolen JS, van Vollenhoven RF, Mease P, Burmester GR, Hiepe F, Khanna D, Nikai E, Coteur G, Schiff M. Certolizumab pegol plus methotrexate provides broad relief from the burden of rheumatoid arthritis: analysis of patient-reported outcomes from the RAPID 2 trial. Ann Rheum Dis. 2011 Jun;70(6):996-1002. doi: 10.1136/ard.2010.143586. Epub 2011 Mar 17. PMID 21415050
- [Result] Hazes JM, Taylor P, Strand V, Purcaru O, Coteur G, Mease P. Physical function improvements and relief from fatigue and pain are associated with increased productivity at work and at home in rheumatoid arthritis patients treated with certolizumab pegol. Rheumatology (Oxford). 2010 Oct;49(10):1900-10. doi: 10.1093/rheumatology/keq109. Epub 2010 Jun 14. PMID 20547658
- [Result] Paul S, Marotte H, Kavanaugh A, Goupille P, Kvien TK, de Longueville M, Mulleman D, Sandborn WJ, Vande Casteele N. Exposure-Response Relationship of Certolizumab Pegol and Achievement of Low Disease Activity and Remission in Patients With Rheumatoid Arthritis. Clin Transl Sci. 2020 Jul;13(4):743-751. doi: 10.1111/cts.12760. Epub 2020 Apr 1. PMID 32100960
- [Derived] Curtis JR, Winthrop K, O'Brien C, Ndlovu MN, de Longueville M, Haraoui B. Use of a baseline risk score to identify the risk of serious infectious events in patients with rheumatoid arthritis during certolizumab pegol treatment. Arthritis Res Ther. 2017 Dec 15;19(1):276. doi: 10.1186/s13075-017-1466-y. PMID 29246162
- [Derived] Smolen JS, van Vollenhoven R, Kavanaugh A, Strand V, Vencovsky J, Schiff M, Landewe R, Haraoui B, Arendt C, Mountian I, Carter D, van der Heijde D. Certolizumab pegol plus methotrexate 5-year results from the rheumatoid arthritis prevention of structural damage (RAPID) 2 randomized controlled trial and long-term extension in rheumatoid arthritis patients. Arthritis Res Ther. 2015 Sep 10;17(1):245. doi: 10.1186/s13075-015-0767-2. PMID 26353833
- [Derived] Combe B, Furst DE, Keystone EC, van der Heijde D, Luijtens K, Ionescu L, Goel N, Emery P. Certolizumab Pegol Efficacy Across Methotrexate Regimens: A Pre-Specified Analysis of Two Phase III Trials. Arthritis Care Res (Hoboken). 2016 Mar;68(3):299-307. doi: 10.1002/acr.22676. PMID 26238672
- [Derived] Kavanaugh A, Smolen JS, Emery P, Purcaru O, Keystone E, Richard L, Strand V, van Vollenhoven RF. Effect of certolizumab pegol with methotrexate on home and work place productivity and social activities in patients with active rheumatoid arthritis. Arthritis Rheum. 2009 Nov 15;61(11):1592-600. doi: 10.1002/art.24828. PMID 19877104